CLINICAL TRIAL: NCT01369602
Title: A Phase 1, Single-Dose, Open-Label Study To Evaluate The Effect Of Renal Impairment On The Pharmacokinetics Of PF-04991532
Brief Title: Study To Evaluate The Effect Of Renal Impairment On The Pharmacokinetics Of PF-04991532
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B2611011
Record Dates: First submitted 2011-06-07; First posted 2011-06-09 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Type 2 Diabetes Mellitus; Healthy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 6-(3-cyclopentyl-2-(4-(trifluoromethyl)-1H-imidazol-1-yl)propanamido)nicotinic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- healthy controls (Experimental): healthy subjects (creatinine clearance > 90 mL/min)
  Interventions: Drug: PF-04991532
- ESRD / severe renal insufficiency (Experimental): Severe (creatinine clearance 15 to 29 mL/min) OR ESRD (creatinine clearnace <15 mL/min OR requiring dialysis)
  Interventions: Drug: PF-04991532
- Moderate renal impairment (Experimental): Moderate (creatinine clearance = 30 to 59 mL/min)
  Interventions: Drug: PF-04991532
- Mild renal impairment (Experimental): Mild (creatinine clearance = 60 to 89 mL/min)
  Interventions: Drug: PF-04991532

INTERVENTIONS:
Drug: PF-04991532 — single dose 300-mg
  Arms: healthy controls
Drug: PF-04991532 — single dose 300-mg
  Arms: ESRD / severe renal insufficiency
Drug: PF-04991532 — single dose 300-mg
  Arms: Moderate renal impairment
Drug: PF-04991532 — single dose 300-mg
  Arms: Mild renal impairment

SUMMARY:
The primary purpose of this study is to evaluate the pharmacokinetics, safety and tolerability of a single oral dose of PF-04991532 in subjects with renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Stable renal function defined as <20% difference between two measurements of serum creatinine obtained on two occasions separated by at least 72 hours to 14 days; the second determination must be obtained within the 28-day period prior to the start of study medication administration. CrCl value at Screening (average of two values obtained within two weeks apart before dosing) will be used for study enrollment.
* Body Mass Index (BMI) of 17.5 to 40 kg/m2; and a total body weight >50 kg (110 lbs).
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of nonhormonal contraception as outlined in this protocol from at least 14 days prior to the first dose of study medication.
* Subjects with recent (within the last 6 months) history of myocardial infarction, unstable angina, coronary revascularization, stroke or transient ischemic attack (TIA).
* Subjects with severe heart failure (New York Heart Association Functional Class IV) at Screening.
* Subjects with acute renal disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUClast) | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 hrs
Maximum observed plasma concentration (Cmax) | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 hrs
Time of maximum observed plasma concentration (Tmax) | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 hrs
Renal Clearance (Clr) | 0 to 24 hours
Amount of drug excreted (Ae) | 0 to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, DeLand, Florida

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2611011&StudyName=Study%20To%20Evaluate%20The%20Effect%20Of%20Renal%20Impairment%20On%20The%20Pharmacokinetics%20Of%20PF-04991532